CLINICAL TRIAL: NCT04016025
Title: Randomized Single-blind Study on the Adherence to Treatment With Topical Methylprednisolone Aceponate (Advantan®) in Different Vehicles (AD-HERE)
Brief Title: A Clinical Study of Adherence to Methylprednisolone Aceponate in Different Carriers
Acronym: AD-HERE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jena University Hospital (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Peter Elsner, Prof. Dr. med. P. Elsner, Head of Dermatology, Principal Investigator, Jena University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZKSJ0119_AD-HERE; 2019-001324-35 (EudraCT Number)
Record Dates: First submitted 2019-06-28; First posted 2019-07-11 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Adherence, Patient; Chronic Eczema
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Intervention Model Description: Randomized single-blind
Who Masked: Care Provider, Investigator
Masking Description: The investigator of the study will not know in which vehicle the enrolled patient will receive the standard therapeutical drug
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cream (Active Comparator): Treatment with topical Methylprednisolone aceponate 0,1% cream (Advantan®) plus Basic care (Bepanthen® Sensiderm)
  Interventions: Behavioral: Adherence to topical standard therapy assessed
- fatty ointment (Active Comparator): Treatment with topical Methylprednisolone aceponate 0,1% fatty ointment (Advantan®) plus Basic care (Bepanthen® Sensiderm)
  Interventions: Behavioral: Adherence to topical standard therapy assessed

INTERVENTIONS:
Behavioral: Adherence to topical standard therapy assessed — Adherence defined as percentage of patients applying at least aimed daily dose

SUMMARY:
Untersuchung der Adhärenz zur topischen Standardtherapie bei Patienten mit chronischem Handekzem in Abhängigkeit von der Galenik

DETAILED DESCRIPTION:
Prospective, randomized, parallel grouped, single-blinded (investigator), monocentric objective assessment of the adherence to the treatment with topical methylprednisolone aceponate (Advantan®) depending on the type of vehicle in patients with hand eczema treated according to the current Guideline.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent has been obtained.
2. Clinical diagnosis of chronic mild-to-moderate hand dermatitis with or without atopic etiology or background (according to IGA: at least mild at Visit 1).
3. Subjects (male or female) aged from 18 to 65 years.
4. In overall good health including well controlled diseases as determined by medical history, physical examination, vital signs and clinical laboratory.
5. Female subjects must be of either:

   * non-childbearing potential, post-menopausal, or have a confirmed clinical history of sterility or,
   * childbearing potential, provided there is a confirmed negative urine pregnancy test prior to exposure, to rule out pregnancy Female subjects of childbearing potential must be willing to use highly effective methods of contraception to avoid causing pregnancy from enrolment and until the last visit (V3).
6. Female subjects must not be breastfeeding.

Exclusion Criteria:

1. females who are pregnant or breast-feeding.
2. Systemic treatment with immunosuppressive drugs, retinoids or corticosteroids within 8 weeks prior to randomization.
3. Phototherapy (PUVA or UVB) on the hands within 4 weeks prior to randomization.
4. Topical applied treatment with immunomodulators (e.g. pimecrolimus or tacrolimus) or corticosteroids on the hands within 2 weeks prior to randomization.
5. Use of other treatment on the hands during the clinical trial except for the use of investigational medicinal product (IMP) and emollient provided by sponsor during the clinical trial.
6. Use of systemic antibiotics or cutaneously applied antibiotics on the hands within 2 weeks prior to randomization.
7. Concurrent skin diseases on the hands and/or integument with acute flare and/or skin lesions within the last 8 weeks.
8. Current diagnosis of eczema on the integument except for the hands.
9. Current diagnosis of exfoliative dermatitis.
10. Current diagnosis of glaucoma or cataract.
11. Significant clinical infection on the hands which requires antibiotic treatment.
12. Known or suspected hypersensitivity to component(s) of the IMP.
13. Subjects with history of an immunocompromising disease (e.g. lymphoma, HIV).
14. Former participation in this clinical trial.
15. Current participation in any other interventional clinical trial.
16. Subjects known or, in the opinion of the investigator, are unlikely to comply with the Clinical Trial Protocol (e.g. alcoholism, drug dependency or psychotic state).
17. Close affiliation with the investigator or other employees of the trial site (e.g. a close relative) or persons working at LEO Pharma A/S or Bayer Consumer Care AG or subject is an employee of sponsor.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2022-03-11 (Actual); Study Completion 2022-04-14 (Actual)

PRIMARY OUTCOMES:
Adherence to treatment | 28 days
  Adherence defined as percentage of patients applying at least aimed daily dose Adherence will be assumed, if
  * truly applicated daily dose is at least 75% of prescribed daily dose and
  * the individual mean number of applications per day is at least 0.85
Measurement 1 | 28 days; visit 1 (day 1)
  Hand surface [cm²]
Measurement 2 | 28 days; visit 1 (day 1), 2 (day 14) and 3 (day 28)
  Weight of topical drug container [mg]
Individual amount of topical drug | 28 days
  - weight of topical drug container [mg] by hand surface [cm²] will be combined to individual amount of topical drug which will as well be the prescribed daily dose
Truly applicated daily dose | 28 days
  - individual amount of topical drug used [mg/cm²] by individual mean number of applications

SECONDARY OUTCOMES:
Change of Hand Eczema | 28 days; visit 1 (day 1), 2 (day 14) and 3 (day 28)
  Hand Eczema Severity Index (HECSI) Score: 0-360 Points (Total HECSI score = Sum (E, I, V, F, S, O) X Ex (Fingertips) + Sum (E, I, V, F, S, O) X Ex (Fingers except tips) + Sum (E, I, V, F, S, O) X Ex (Palm of hands) + Sum (E, I, V, F, S, O) X Ex (Back of hands) + Sum (E, I, V, F, S, O) X Ex (Wrists))
Change of Hand Eczema | 28 days; visit 1 (day 1), 2 (day 14) and 3 (day 28)
  Investigator's global Assessment (IGA) Score: 0-4 Points (0=Clear, 1=Almost clear, 2=Mild, 3=Moderate, 4=Severe)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Elsner, Prof. Dr. med., Principal Investigator — University hospital Jena
Locations (1):
- Jena University Hospital, Jena, Thuringia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Diepgen TL, Andersen KE, Chosidow O, Coenraads PJ, Elsner P, English J, Fartasch M, Gimenez-Arnau A, Nixon R, Sasseville D, Agner T. Guidelines for diagnosis, prevention and treatment of hand eczema. J Dtsch Dermatol Ges. 2015 Jan;13(1):e1-22. doi: 10.1111/ddg.12510_1. PMID 25763418
- [Background] Torrelo A. Methylprednisolone aceponate for atopic dermatitis. Int J Dermatol. 2017 Jun;56(6):691-697. doi: 10.1111/ijd.13485. Epub 2017 Mar 4. PMID 28258632
- [Background] Schliemann S, Petri M, Elsner P. How much skin protection cream is actually applied in the workplace? Determination of dose per skin surface area in nurses. Contact Dermatitis. 2012 Oct;67(4):229-33. doi: 10.1111/j.1600-0536.2012.02119.x. Epub 2012 Jun 18. PMID 22709142
- [Background] Lee JY, Choi JW, Kim H. Determination of hand surface area by sex and body shape using alginate. J Physiol Anthropol. 2007 Jun;26(4):475-83. doi: 10.2114/jpa2.26.475. PMID 17704626
- [Background] Gray R, Wykes T, Gournay K. From compliance to concordance: a review of the literature on interventions to enhance compliance with antipsychotic medication. J Psychiatr Ment Health Nurs. 2002 Jun;9(3):277-84. doi: 10.1046/j.1365-2850.2002.00474.x. PMID 12060371
- [Background] Ofenloch RF, Weisshaar E, Dumke AK, Molin S, Diepgen TL, Apfelbacher C. The Quality of Life in Hand Eczema Questionnaire (QOLHEQ): validation of the German version of a new disease-specific measure of quality of life for patients with hand eczema. Br J Dermatol. 2014 Aug;171(2):304-12. doi: 10.1111/bjd.12819. Epub 2014 Jun 18. PMID 24397866
- [Background] Agner T, Jungersted JM, Coenraads PJ, Diepgen T. Comparison of four methods for assessment of severity of hand eczema. Contact Dermatitis. 2013 Aug;69(2):107-11. doi: 10.1111/cod.12039. PMID 23869730
- [Background] Ruzicka T, Lynde CW, Jemec GB, Diepgen T, Berth-Jones J, Coenraads PJ, Kaszuba A, Bissonnette R, Varjonen E, Hollo P, Cambazard F, Lahfa M, Elsner P, Nyberg F, Svensson A, Brown TC, Harsch M, Maares J. Efficacy and safety of oral alitretinoin (9-cis retinoic acid) in patients with severe chronic hand eczema refractory to topical corticosteroids: results of a randomized, double-blind, placebo-controlled, multicentre trial. Br J Dermatol. 2008 Apr;158(4):808-17. doi: 10.1111/j.1365-2133.2008.08487.x. Epub 2008 Feb 21. PMID 18294310
- [Background] Reich A, Chatzigeorkidis E, Zeidler C, Osada N, Furue M, Takamori K, Ebata T, Augustin M, Szepietowski JC, Stander S. Tailoring the Cut-off Values of the Visual Analogue Scale and Numeric Rating Scale in Itch Assessment. Acta Derm Venereol. 2017 Jun 9;97(6):759-760. doi: 10.2340/00015555-2642. No abstract available. PMID 28224165